CLINICAL TRIAL: NCT01005082
Title: Calcium Nephrolithiasis: Clinical Characteristics and Nutritional Determinants
Brief Title: Low Salt Diet in Idiopathic Hypercalciuria
Acronym: LOSALT01
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Parma (Other)
Collaborators: Università Vita-Salute San Raffaele (Other); University of Milan (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: University of Parma, University of Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIN2002062925
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Hypercalciuria
Keywords: Low salt diet, idiopathic hypercalciuria, calcium stone formers; Calcium stone formers with idiopathic hypercalciuria
MeSH Terms: conditions — Hypercalciuria | interventions — Diet, Sodium-Restricted; Water

ARMS (2):
- Low salt diet plus water therapy (Experimental)
  Interventions: Behavioral: Low salt diet
- water therapy alone (Active Comparator)
  Interventions: Behavioral: Water therapy alone

INTERVENTIONS:
Behavioral: Low salt diet
  Arms: Low salt diet plus water therapy
Behavioral: Water therapy alone
  Arms: water therapy alone

SUMMARY:
Randomized clinical trial comparing water therapy plus low-salt diet to water therapy alone in patients affected by idiopathic calcium nephrolithiasis.

Treatment duration: three months Primary end-point: correction of hypercalciuria Main inclusion criteria: calcium stone formers with idiopathic hypercalciuria, with at least one stone expelled and analyzed by infrared spectrophotometry; presence of hypercalciuria (>300 mg/day in males and >200 mg/day in females); 18-65 years.

Main exclusion criteria: primary hyperparathyroidism, primary hyperoxaluria, enteric hyperoxaluria, bowel resection, inflammatory bowel disease, renal tubular acidosis, sarcoidosis, sponge kidney, hyperthyroidism, use of hypercalciuric drugs such as Vitamin D, acetazolamide, anti-epileptic drugs

ELIGIBILITY:
Main inclusion criteria:

* idiopathic calcium stone formers, with at least one stone expelled and analyzed by infrared spectrophotometry; presence of hypercalciuria (>300 mg/day in males and 20 mg/day in females);
* 18-65 years.

Main exclusion criteria:

* primary hyperparathyroidism,
* primary hyperoxaluria,
* enteric hyperoxaluria,
* bowel resection,
* inflammatory bowel disease,
* renal tubular acidosis,
* sarcoidosis, sponge kidney,
* hyperthyroidism,
* use of hypercalciuric drugs such as Vitamin D,
* acetazolamide,
* anti-epileptic drugs

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2005-01; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Normalization of urinary calcium levels

SECONDARY OUTCOMES:
Change in urinary stone risk factors (e.g. urinary calcium, oxalate and sodium excretion); blood pressure reduction

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Parma, Italy

REFERENCES:
- [Background] Borghi L, Schianchi T, Meschi T, Guerra A, Allegri F, Maggiore U, Novarini A. Comparison of two diets for the prevention of recurrent stones in idiopathic hypercalciuria. N Engl J Med. 2002 Jan 10;346(2):77-84. doi: 10.1056/NEJMoa010369. PMID 11784873
- [Derived] Nouvenne A, Meschi T, Prati B, Guerra A, Allegri F, Vezzoli G, Soldati L, Gambaro G, Maggiore U, Borghi L. Effects of a low-salt diet on idiopathic hypercalciuria in calcium-oxalate stone formers: a 3-mo randomized controlled trial. Am J Clin Nutr. 2010 Mar;91(3):565-70. doi: 10.3945/ajcn.2009.28614. Epub 2009 Dec 30. PMID 20042524